CLINICAL TRIAL: NCT00002369
Title: An Open Label, Randomized, Comparative Study of Zerit (d4T) + Epivir (3TC) + Crixivan Versus Retrovir (AZT) + Epivir (3TC) + Crixivan in HIV-Infected, Antiretroviral Naive Subjects With CD4 Cell Counts of 200 - 700 Cells/mm3 and HIV RNA Baseline Copy Number of >= 10,000 Copies/ml
Brief Title: A Comparison of Epivir Plus Crixivan Combined With Zerit or Retrovir in HIV-Infected Patients Who Have Never Taken Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 260A; BMS 001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; Stavudine; HIV Protease Inhibitors; CD4 Lymphocyte Count; Lamivudine; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
To evaluate the tolerance, and comparative virologic and immunologic effects of the two combination regimens.

DETAILED DESCRIPTION:
100 patients will be randomized to receive Zerit (Stavudine) + Epivir (Lamivudine) + Crixivan (Indinavir) and 100 patients will be randomized to receive Retrovir (Zidovudine) + Epivir (Lamivudine) + Crixivan (Indinavir).

Patients will be treated for 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 cell count of 200 - 700 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

AIDS defining condition within 1 month of study entry.

Prior Medication:

Excluded:

Patients with any history of antiretroviral therapy treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - HIV Clinical Research Ctr, Fort Lauderdale, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Advance Clinical Research, Atlanta, Georgia
  - Louisiana State Univ Med Ctr / HIV Outpatient Clinic, New Orleans, Louisiana
  - Boston Univ Med Ctr Hosp / Evans - 556, Boston, Massachusetts
  - Community Research Initiative of New England, Brookline, Massachusetts
  - Washington Univ School of Medicine, St Louis, Missouri
  - Blackstock Family Health Ctr, Austin, Texas
- Puerto Rico (2):
  - Hosp Regional de Ponce - Area Vieja, Ponce
  - San Juan AIDS Program, Santurce